CLINICAL TRIAL: NCT01479439
Title: A Phase II Trial of Losartan to Reverse Sickle Nephropathy
Brief Title: Losartan to Reverse Sickle Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-3070
Record Dates: First submitted 2011-11-16; First posted 2011-11-24 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Nephropathy; Sickle Cell Anemia
MeSH Terms: conditions — Kidney Diseases; Anemia, Sickle Cell | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sickle cell disease (Experimental): The purpose of this research study is to see if losartan can help reduce or reverse damage done to the kidneys of children and adults with Sickle Cell Anemia (SCA) and Sickle Beta-zero (HbSβ0) Thalassemia.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — Form: suspension, tablet. Dosage & frequency: age 6-16 = 0.7mg/kg once daily; age >16 = 50mg once daily. Duration: 6 months

SUMMARY:
Sickle cell disease causes kidney damage with increasing age, leading to chronic kidney disease and renal failure in nearly one third of patients with sickle cell disease. Currently, there is no treatment for sickle cell related kidney disease.

DETAILED DESCRIPTION:
The purpose of this research study is to see if losartan can help reduce or reverse damage done to the kidneys of children and adults with Sickle Cell Anemia (SCA) and Sickle Beta-zero (HbSβ0) Thalassemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥6 years of age; for no albuminuria (NoA) group age is ≥ 6 years and <21 years of age
2. Diagnosis of hemoglobin SS disease or Sβ0 thalassemia by hemoglobin electrophoresis and/or β-globin gene mapping.
3. Urine osmolality <700 mOsm (milliosmoles) on first morning urine
4. Written informed consent (and assent, where applicable)
5. Documented urine albumin to creatinine ratio (UACR) showing either

   * NoA: UACR <30mg/g creatinine on a first morning urine
   * MiA: UACR 30-300 mg/g creatinine on a first morning urine or
   * MaA: UACR >300 mg/g creatinine on a first morning urine sample
6. A documented negative serum pregnancy test for females with child bearing potential or greater than 10 years of age within (prior to) 7 days of starting the study medication.
7. Subjects with child-bearing potential must be willing to use a medically accepted form of contraception throughout the study.
8. Patients on hydroxyurea (HU) who are on a stable (not changing) dose of HU for three months prior to study entry.

Exclusion Criteria:

1. Patients with Hb SC, SD, Sβ+thal, SE and other sickle hemoglobinopathies, and sickle trait (AS).
2. Pregnant or lactating females, or females of child-bearing potential that are unable to use a medically accepted form of contraception throughout the study.
3. Urine creatinine clearance (Clcr) <60 mL/minute/1.73 m2
4. Gross (not microscopic) hematuria. If hematuria has resolved for 2 weeks or more, patients will be eligible.
5. Hyperkalemia (K≥5.5) at baseline despite a low potassium diet
6. Concurrent condition that predisposes to nephropathy, such as lupus, diabetes, and hypertension, not controlled with medications..
7. On a renin-angiotensin pathway inhibitor (e.g., captopril, lisinopril, Losartan, valsartan, etc) for the last two weeks prior to enrollment.
8. Hypersensitivity to Angiotensin II receptor blockers such as losartan, valsartan, telmisartan.
9. Patients on red cell apheresis or ongoing aggressive chronic transfusions (one or more a month with a goal of HbS < 30%). Patients receiving a simple transfusion for symptoms during acute event will be eligible, but if they receive a partial or full exchange transfusion during an acute event, then they will only be eligible after 90 days.
10. Hepatic dysfunction defined as ALT (alanine aminotransferase) or direct bilirubin > 3-times upper limit of normal (ULN).
11. Chronic therapy with NSAIDS or Cox2 inhibitors
12. On another interventional trial. May be eligible two weeks after completion of another interventional study.
13. Any condition that interferes with the ability of the patient to understand or comply with the treatment plan and follow up.
14. A serious mental or physical illness or a major disease (cardiac, renal, hepatic, neurological, endocrine, metabolic, pulmonary function or psychiatric), which in the opinion of the investigator would compromise participation in the study.
15. Unable to take oral medications.
16. HIV confirmed positive.
17. Chronic therapy with steroids. May be eligible after three weeks of completing steroid therapy.
18. Patients on lithium will be excluded

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Punam Malik, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (9):
- United States (9):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - NHLBI, Bethesda, Maryland
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Texas Southwestern, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Quinn CT, Saraf SL, Gordeuk VR, Fitzhugh CD, Creary SE, Bodas P, George A, Raj AB, Nero AC, Terrell CE, McCord L, Lane A, Ackerman HC, Yang Y, Niss O, Taylor MD, Devarajan P, Malik P. Losartan for the nephropathy of sickle cell anemia: A phase-2, multicenter trial. Am J Hematol. 2017 Sep;92(9):E520-E528. doi: 10.1002/ajh.24810. Epub 2017 Jul 19. PMID 28589652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, phase 2, open-label study of losartan for sickle cell nephropathy. Participants were enrolled at nine centers in the United States between 2012 and 2015.
Pre-assignment Details: Concomitant treatment with hydroxyurea was allowed, but the dose must have been stable in the 3 months preceding enrollment. Participants were allocated to three pre-specified groups defined by baseline urinary albumin-to-creatinine ratio (UACR).
Groups:
- Losartan - No Albuminuria: Baseline urinary albumin-to-creatinine ratio (UACR) <30 mg/g.
  All participants in this study in all arms were treated with losartan using the same dosing regimen. Study arms are only differentiated by baseline UACR.
- Losartan - Microalbuminuria: Baseline urinary albumin-to-creatinine ratio (UACR) 30-300 mg/g.
  All participants in this study in all arms were treated with losartan using the same dosing regimen. Study arms are only differentiated by baseline UACR.
- Losartan - Macroalbuminuria: Baseline urinary albumin-to-creatinine ratio (UACR) >300 mg/g.
  All participants in this study in all arms were treated with losartan using the same dosing regimen. Study arms are only differentiated by baseline UACR.
Period: Overall Study
Arm/Group | Losartan - No Albuminuria | Losartan - Microalbuminuria | Losartan - Macroalbuminuria
Started | 15 | 13 | 8
Completed | 14 | 12 | 6
Not Completed | 1 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan - No Albuminuria | Losartan - Microalbuminuria | Losartan - Macroalbuminuria | Total
Number analyzed (Participants) | 14 | 12 | 6 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 4 | 1 | 14
  Between 18 and 65 years | 5 | 8 | 5 | 18
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (4.9) | 28.6 (16.6) | 38.8 (18.5) | 24.4 (88.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 4 | 18
  Male | 8 | 4 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 12 | 6 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 12 | 6 | 32
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 6 | 32
Urinary albumin-to-creatinine ratio (UACR) (mg/g) [Mean (Standard Deviation); unit: mg/g] — The ratio of urinary albumin concentration (in mg) to urinary creatinine concentration (in g).
  mg/g | 8.5 (4.9) | 121 (86.6) | 815 (335.6) | 202 (333.8)
Creatinine clearance by 24h Urine Collection [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 146 (228) | 172 (204) | 108 (46.5) | 150 (56.5)

OUTCOME MEASURES:

1. Primary Outcome: Categorical Change in Urinary Albumin-to-creatinine Ratio (UACR) From Baseline
Description: Number of participants who have a ≥25% reduction in urinary albumin-to-creatinine ratio (UACR) from baseline to 6 months. This is a categorical outcome (yes/no).
  We hypothesized and pre-specified that ≥30% of the subjects in the microalbuminuria group would meet this outcome.
Time Frame: Baseline and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan - No Albuminuria | Losartan - Microalbuminuria | Losartan - Macroalbuminuria
Number analyzed (Participants) | 14 | 12 | 6
Participants | 1 | 7 | 5

2. Secondary Outcome: Change in UACR
Description: Fold-change in UACR from baseline
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: Fold-change
Groups:
- No Albuminuria (NoA): Baseline urinary albumin-to-creatinine ratio (UACR) <30 mg/g
- Microalbuminuria (MicroA): Baseline urinary albumin-to-creatinine ratio (UACR) 30-300 mg/g
- Macroalbuminuria: Baseline urinary albumin-to-creatinine ratio (UACR) >300 mg/g
Arm/Group | No Albuminuria (NoA) | Microalbuminuria (MicroA) | Macroalbuminuria
Number analyzed (Participants) | 14 | 12 | 6
Fold-change | 0.08 [-0.07 to 1.06] | -0.46 [-0.75 to 2.53] | -0.74 [-0.91 to -0.17]

3. Secondary Outcome: Change in Creatinine Clearance
Description: Fold-change in creatinine clearance by 24h urine collection (GFR-CrCl) from baseline
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: Fold-change
Arm/Group | No Albuminuria (NoA) | Microalbuminuria (MicroA) | Macroalbuminuria
Number analyzed (Participants) | 14 | 12 | 6
Fold-change | 0.06 [-0.10 to 0.44] | 0.12 [-0.34 to 0.26] | 0.05 [-0.01 to 0.33]

ADVERSE EVENTS:
Arm/Group | No Albuminuria (NoA) | Microalbuminuria (MicroA) | Macroalbuminuria
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 0/14 | 1/12 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Albuminuria (NoA) (N=14) | Microalbuminuria (MicroA) (N=12) | Macroalbuminuria (N=6)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Increase in serum creatinine >50% from baseline (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Decline in GFR >25% from baseline (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
We cannot conclude from this small phase 2 study that losartan is efficacious for sickle cell nephropathy. Rather, the data generated from this study will inform the design of a phase-3 randomized trial to determine its efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No